CLINICAL TRIAL: NCT07206199
Title: Virtual Reality Exposure Therapy in Patients With Obsessive-Compulsive Disorder: A Randomized Controlled Trial in Outpatients
Brief Title: Virtual Reality Exposure Therapy for Obsessive-Compulsive Disorder: Outpatients Trial
Acronym: OCD-VRET2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health, Czech Republic (Other)
Responsible Party: Principal Investigator, Iveta Fajnerová, Supervisor, National Institute of Mental Health, Czech Republic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU23-04-00402-Study2
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Obsessive-compulsive Disorder
Keywords: Obsessive-compulsive disorder; virtual reality; Virtual reality exposure therapy; within-subject design; Outpatients
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Implosive Therapy; Waiting Lists

STUDY DESIGN:
Intervention Model Description: Within-subject design. Waiting list period followed by active treatment period of the same length (5 weeks).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Within-subject comparison of a waiting list condition with exposure therapy in VR (Experimental): Patients first complete informed consent and baseline questionnaires and are placed on a waiting list for five weeks. After this period, they are reassigned to the active group, which receives five sessions of exposure therapy in virtual reality over a subsequent five-week period. The treatment effect will be evaluated using pre/post assessments, as well as monitoring adherence to exposure and response prevention assignments.
  Interventions: Behavioral: exposure therapy in virtual reality; Other: Wait list

INTERVENTIONS:
Behavioral: exposure therapy in virtual reality — Participants complete five 30-40-minute sessions of exposure therapy administered via a virtual reality headset once a week. The exposure involves exposure to various symptom-provoking scenarios in the virtual house environment. Scenarios can be adjusted to distinct OCD dimensions: contamination/cleaning, fear-of-harm/checking symmetry/ordering, and also to symptoms of hoarding. Stimuli can be also freely combined across different dimensions, so that the scenarios fit the individual needs.
Other: Wait list — The patients are assigned to a waitlist period for 5 weeks. During this period they are not allowed to change any treatment (phramacotherapy and/or psychoterapy as usual) started prior to the trial.

SUMMARY:
The aim of this study is to evaluate the efficacy of virtual reality exposure therapy (VRET) as a treatment for obsessive-compulsive disorder (OCD). This study focuses on patients receiving treatment in outpatient psychiatry or clinical psychology settings, utilizing a within-subject design for comparison. Patients first complete informed consent and baseline questionnaires and are placed on a waiting list for five weeks. After this period, they are reassigned to the active (experimental) group, which will receive five sessions of exposure therapy in virtual reality over a subsequent five-week period. The treatment effect will be evaluated using pre/post assessments, as well as monitoring adherence to exposure and response prevention assignments.

DETAILED DESCRIPTION:
The virtual environment of so called "OCD house" is used as a tool for the therapy. Immersive VR glasses Meta Quest 2 are used to visualize the environment.

During exposure therapy, relevant virtual stimuli can be freely combined involving common objects and situations in the home that may trigger OCD symptoms and hoarding. Target stimuli (VR elements) are divided into several sets corresponding to OCD subtypes. During the session, the therapist can modify the level of difficulty via four standardized levels according to the individual needs of clients.

The therapeutic application enables direct interaction with stimuli in the environment of the virtual house and garden, thanks to hand tracking. The hand tracking and hand gestures are used also to control the movement in the environment by the patients, but direct head and body rotations and small movements are enabled by the VR headset. The psychotherapist can follow the patient actions and control the settings of the environment (e.g.selection of relevant stimuli, level of difficulty) using a streaming app on the tablet or a mobile phone and advise the patient where necessary. The level of difficulty is gradually increased during the progress of the therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OCD (F42) using currently valid DSM-V and ICD-11
* Fluent in Czech

Exclusion Criteria:

* Any other psychiatric, neurological and serious somatic illness
* Substance abuse
* Psychotropic medication (e.g. benzodiazepines) except antidepressants, antipsychotic medication and hypnotics.
* Contradictions to using a virtual reality (e.g., epilepsy, balance problems)
* Pregnancy
* Cardiostimulator and mental implants

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
The Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) self report version | Applied repeatedly: 1) Before the assignment to the waitlist condition, 2) After the waitlist period = Before the start of the first VRET therapy session, 3) After the last VRET session and 4) Follow-up 3 months after the last therapy session.
  The Y-BOCS is a 19-item scale assessing the severity of obsessive-compulsive symptoms. Raw score range from 0 to 40, where 0 = no symptoms and 40 = very severe symptoms with highly impaired daily functioning.
The Beck Depression Inventory | Applied repeatedly: 1) Before the assignment to the waitlist condition, 2) After the waitlist period = Before the start of the first VRET therapy session, 3) After the last VRET session and 4) Follow-up 3 months after the last therapy session.
  The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression.
Beck Anxiety Inventory (BAI) | Applied repeatedly: 1) Before the assignment to the waitlist condition, 2) After the waitlist period = Before the start of the first VRET therapy session, 3) After the last VRET session and 4) Follow-up 3 months after the last therapy session.
  BAI is an inventory of anxiety symptoms with 18 items rated on a 5-point Likert scale (0-4). Score range from 0 to 72, with higher scores indicating more severe anxiety symptoms.
Hierarchy of fears | Applied repeatedly: 1) Before the assignment to the waitlist condition, 2) After the waitlist period = Before the start of the first VRET therapy session, 3) After the last VRET session and 4) Follow-up 3 months after the last therapy session.
  Patients describe and rate their most feared situations or stimuli on a 10-point scale (1-10).
The Spielberger State-Trait Anxiety Inventory-X2 (STAI-X2) | Applied repeatedly: 1) Before the assignment to the waitlist, 2) After the waitlist period = Before the start of the first VRET therapy session, 3) After the last VRET session and 4) Follow-up 3 months after the last therapy session
  The Spielberger State-Trait Anxiety Inventory-X2 (STAI-X2) is used to measure self-reported symptoms of trait anxiety with higher score indicating higher anxiety levels (score range 20-80).

SECONDARY OUTCOMES:
Subjective Units of Distress Scale (SUDS) | During In-Sessions: week 1-5 of experimental VRET condition
  The SUDS is a visual analog scale in which the participant rates his/her anxiety/discomfort based on a range between 1 (no anxiety/discomfort) and 10 (very severe anxiety/discomfort).
Adherence to exposures | Before In-Sessions: week 1-5 of experimental VRET condition
  Four questions aimed at gathering information about how patients managed to perform exposures during the past week and to what extent the skills acquired during the VR exposure therapy were useful.
The Igroup Presence Questionnaire (IPQ) | Immediately after the first session of VR exposure therapy.
  The scale includes 3 subscales SP (spatial presence), INV (involvement) and REAL (experienced realism) with score range 0-7. Higher scores indication higher sense of presence. This measure might be positivelly associated with positive outcome.
Simulator Sickness Questionnaire (SSQ) | Immediately after the first session of VR exposure therapy.
  The scale evaluates cybersickness symptoms in three subscales: nausea (N), oculomotor disturbance (O), disorientation (D). Total simulator sickness raw score 0-48 (adjusted total score 0-180). Higher scores on each scale indicatestronger perceptions of the underlying sickness symptoms and aretherefore undesired. This measure might be negatively associated with positive outcome and sense of presence.

CONTACTS AND LOCATIONS:
Overall Officials: Iveta Hocko Fajnerová, Ph.D., Study Director — National Institute of Mental Health (NIMH); Pavla Stopková, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- Nationa Institute of Mental Health, Klecany, Česká Republika, Czechia

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the publication of results
Supporting Information: Study Protocol, SAP
Time Frame: After the publication of study data.
Access Criteria: The anonymized preprocessed behavioral data will be shared using an institutional open access or journal repository. Additional raw data access requests will be reviewed using an online form. Requestors will be required to sign a data access agreement.

REFERENCES:
- See also: Description and illustration images of the software used in the study. — https://ocddum.cz/en